CLINICAL TRIAL: NCT07169669
Title: Multicentre Longitudinal Study of Bone Mineralisation Characteristics in Marfan Syndrome and Ehlers-Danlos Syndrome
Acronym: BONE
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: BONE
Record Dates: First submitted 2025-09-04; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Marfan Syndrome; Ehlers-Danlos Syndrome (EDS); Mineral Density
MeSH Terms: conditions — Marfan Syndrome; Ehlers-Danlos Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Marfan group: Adult and paediatric subjects with Marfan syndrome referred to the Centre for Cardiovascular Genetic of IRCCS Policlinico San Donato
- Ehlers Danlos group: Adult and paediatric subjects with Ehlers Danlos Syndrome referred to the Centre for CardioVascular Genetics of IRCCS Policlinico San Donato and the Reference Centre for Ehlers-Danlos Syndromes Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico

SUMMARY:
The general objective of this research is to evaluate the characteristics of bone mineralisation in patients with Marfan syndrome or Ehlers-Danlos syndrome on a large case series.

In particular we intend to obtain data regarding the characteristics of bone mineralisation, as well as their variation over time and the relationships existing with other clinical-anamnestic parameters, in patients with Marfan syndrome or Ehlers-Danlos syndrome by retrospectively analysing (data already collected for normal clinical practice and already available at the hospital) the case history of the Cardiovascular genetic center at IRCCS Policlinico San Donato and the related Computerized Bone Mineralometry (MOC) examinations performed at the Radiology Service of the same hospital between 1 September 2019 and 31 December 2022.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Marfan syndrome and Ehlers-Danlos syndrome according to the revised reference criteria belonging to the Cardiovascular genetic center at IRCCS Policlinico San Donato and the Reference Centre for Ehlers-Danlos Syndromes Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico;
* Adult and paediatric subjects who have performed at least one Bone Mineral Densitometry within the observation period of the study.

Exclusion Criteria:

* Presence of prostheses in the spinal column;
* Presence of prostheses in the coxofemoral joint;
* Oncological bone diseases reported in history.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Marfan syndrome is a rare connective tissue disease with autosomal dominant transmission, characterised by altered production of the glycoprotein fibrillin-1 (FBN1), resulting from mutations in the gene encoding it.The complications most associated with the risk of mortality and morbidity are those affecting the cardiovascular system and those affecting the musculoskeletal system (spinal changes and chest deformities).
  Ehlers-Danlos syndrome has an estimated prevalence of 1:5000 individuals and presents a pathological phenotype affecting the connective tissues that support the integumentary, skeletal, cardiovascular, and other organs and tissues. As in Marfan syndrome, marked alterations in the skeletal system (spine, thorax) and, in the vascular forms, a high risk of aneurysms and aortic and/or small and medium artery dissection, are found in those with Ehlers-Danlos syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective 1 | Between 1 September 2019 and 31 January 2025.
  To retrospectively evaluate the percentage of subjects with fractures in subjects with Marfan syndrome and Ehlers Danlos syndrome who performed at least one Bone Mineral Densitometry in the period between 1 September 2019 and 31 January 2025.

SECONDARY OUTCOMES:
Objective 2 | Between 1 September 2019 and 31 January 2025.
  Identifying patients with osteoporosis with T-score values below -2.5 SD and z-score values ≤ -2 SD in the paediatric population.
Objective 3 | Between 1 September 2019 and 31 January 2025.
  Identify patients with osteopenia with T scores between -1 and -2.5 SD
Objective 4 | Between 1 September 2019 and 31 January 2025.
  Identify adult patients with TBS values
  * TBS values ≤ 1200 (degraded micro-architecture);
  * TBS values between 1349 - 1201 (partially degraded micro-architecture).